CLINICAL TRIAL: NCT03702556
Title: The Representation of the Breast on the Somatosensory Cortex After Autologous Breast Reconstruction Using 7 Tesla Functional MRI.
Brief Title: Functional MRI Study Reconstructed Breasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL67696.068.18
Record Dates: First submitted 2018-10-07; First posted 2018-10-11 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mastectomy without breast reconstruction (Active Comparator): Functional MRI scan of the somatosensory cortex while the breast skin is stimulated by piezo-stimulators.
  Interventions: Device: MRI scan
- Breast reconstruction with nerve (Active Comparator): Functional MRI scan of the somatosensory cortex while the breast skin is stimulated by piezo-stimulators.
  Interventions: Device: MRI scan
- Breast reconstruction without nerve (Active Comparator): Functional MRI scan of the somatosensory cortex while the breast skin is stimulated by piezo-stimulators.
  Interventions: Device: MRI scan

INTERVENTIONS:
Device: MRI scan — 7.0 tesla functional MRI scan

SUMMARY:
Rationale: To study the effects of mastectomy and autologous breast reconstruction on the sensation of the (reconstructed) breast, not only the peripheral reinnervation of the breast should be studied, but also the changes that take place in the somatosensory cortex. Now that the region of interest in the brain and the somatotopy of the non-operated breast are known, studies with patients who underwent mastectomy and breast reconstruction are the next step to understand the neuroplasticity of the brain following breast surgery.

Objective: To study the neuroplasticity of the brain after mastectomy and breast reconstructive surgery by assessing the somatotopy of the breast on the somatosensory cortex of patients who underwent either breast reconstruction with and without nerve restoration or mastectomy without breast reconstruction.

Study design: A single center imaging study carried out in Maastricht University Medical Center.

Study population: A total of 30 female breast cancer patients who underwent a unilateral mastectomy without breast reconstruction or a mastectomy followed by a unilateral autologous breast reconstruction with a deep inferior epigastric artery perforator (DIEP) flap will be included in this study. Three groups of patients will be selected and compared: ten patients who underwent a mastectomy without breast reconstruction, ten patients who underwent a DIEP flap breast reconstruction with sensory nerve restoration of the flap and ten patients who underwent a DIEP flap without nerve restoration.

Intervention: Every subject will undergo a single functional MRI scan in a 7 Tesla MRI scan at least six months after the operation. A scanning session takes approximately 75 minutes. During the scan, piezo-electric stimulators are applied to both the reconstructed and non-operated breast in a fixed pattern. These stimulators stimulate the skin and sensory nerves of the breast and nipple-areola complex in a random sequence.

Main study parameters: The hemodynamic response after stimulation of the skin of the breast and nipple-areola complex, representing neuronal activity in that region, is measured. Within the somatosensory cortex (S1 and S2), the temporo-spatial brain activity patterns after the various stimulation conditions are assessed, and the representation of the breast on the somatosensory cortex is mapped.

ELIGIBILITY:
Inclusion Criteria:

* Female over 18 years old
* Unilateral mastectomy without breast reconstruction
* Unilateral mastectomy with DIEP flap breast reconstruction (with or without sensory nerve restoration)
* At least six months after the operation
* Informed consent

Exclusion Criteria:

* Bilateral mastectomy / breast reconstruction
* Previous surgery, disease or treatment of the contralateral breast
* Active disease / metastasis
* Previous radiation therapy on the chest or axilla
* Diseases associated with neuropathy (e.g. diabetes mellitus)
* Previous brain surgery
* Previous allergic reactions to adhesives or plasters
* Any MRI exclusion criteria:

  * No piercings or other iron materials (except a metal brace behind front teeth)
  * Claustrophobia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
The neuroplasticity of the brain after breast reconstruction | 75 minutes
  Changes in the blood oxygen level dependent (BOLD) contrast as a function of vibrotactile stimulation of the breast and nipple-areola complex will be measured. Changes will be analysed using multi-voxel pattern analysis to localize the different parts of the breast in the somatosensory cortex.

SECONDARY OUTCOMES:
Differences in the somatotopy between patients who underwent a breast reconstruction with nerve restoration compared to patients who underwent breast reconstruction without nerve restoration. | 75 minutes
  Differences between groups in somatotopy of the breast in the somatosensory cortex will be assessed.
Differences in the somatotopy between patients who underwent mastectomy without breast reconstruction compared to patients who underwent breast reconstruction. | 75 minutes
  Differences between groups in somatotopy of the breast in the somatosensory cortex will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: René Van der Hulst, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided